CLINICAL TRIAL: NCT04708873
Title: Effect of High Intensity Aerobic & Resistance Interval Training on Body Composition, Visceral Adiposity and Myocardial Function in Overweight and Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/13
Record Dates: First submitted 2021-01-01; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to Interventional Group A (High intensity aerobic & resistance interval training) or Interventional Group B/ Control Group (Moderate intesity continuous training) for the whole duration of the study.
Who Masked: Participant
Masking Description: It will be a single blinded study. Only the participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training Group (Experimental): Participants in this group will initially undergo continuous aerobic training to achieve a baseline fitness level, after which HIIT and resistance training will be employed. Warm-up period will be followed by 4 bouts of 4-minute interval treadmill running and stationary bike cycling at 80-95% of the measured HR reserve, interspersed with active recovery phase at 55-70% HRR. After this resistance exercises will be performed in a circuit fashion for strengthening the upper limbs, lower limbs and trunk. The session will be ended with a 5-7 minute cool-down period
  Interventions: Other: High intensity interval training
- Moderate Intensity Continuous Training Group (Active Comparator): Participants in this group will also initially undergo continuous aerobic training to achieve a baseline fitness level, after which the intensity will be increased to moderate continuous training achieving 55-70% of HRR. Every session will be preceded by appropriate warm-up and end with cool down.
  Interventions: Other: Moderate Intensity Continuous Training

INTERVENTIONS:
Other: High intensity interval training — 4x4 min intervals of high intensity treadmill running (80-95% of HRR, RPE 7-10 on Borg's category ratio scale of perceived exertion) interspersed with active recovery (slow jogging or fast walking at 50-70% HRR). HIIT-Resistance exercises 2 sessions per week, RPE 5 (hard) 6-8 RM, 1-3 sets of as many repetitions as possible in 60 seconds, active recovery 20-60 seconds b/w exercises,
  Arms: High Intensity Interval Training Group
Other: Moderate Intensity Continuous Training — Moderate intensity continuous Aerobic exercises (Stationary cycling for 15-20 min followed by treadmill walking for 15-20 min) at 55-70% 55-70% of HRR, RPE 3-4 on Borg's category ratio scale of perceived exertion. The session will be preceded by 5-7 minute warm-up & 7-10 min cool-down.
  Arms: Moderate Intensity Continuous Training Group

SUMMARY:
The obesity epidemic, predisposing to cardio-metabolic diseases, has increased two-folds over the last decade with a global alarming cost of obesity-associated illnesses, thus representing a grave peril for the survival of public health care systems. It is need of the time to develop evidence-based, time-efficient and cost-effective strategies to prevent and manage obesity. This study would compare the effects of 2 types of exercise regimes providing data on their beneficial effects on body composition and myocardial function along with reducing the central adiposity. This study may also be used as a novel intervention strategy for primary prevention of cardiovascular and metabolic diseases by modification of a major risk factor i.e. obesity in Pakistani population, consequently reducing the burden of morbidity and mortality from cardiometabolic diseases.

DETAILED DESCRIPTION:
Obesity is one of the major public health issues of this century. Over the last decade, the prevalence of obesity has increased globally, making it an emerging epidemic and threatening the survival of health care systems. Obesity has long been recognized as the major factor predisposing to cardio-metabolic diseases.The positive role of structured exercise for reducing the mortality and morbidity rates of obese and sedentary adults is well established. But exercise engagement is seen to be quite low in obese adults mainly due to lack of time and non-adherence to exercise training programs. Current trends are now focusing towards another type of exercise regime known as high intensity interval training (HIIT), which is composed of repetitive short to long (< 45 sec to 4 min) bouts of high intensity exercise alternating with rest or recovery periods. Resistance training can also stimulate changes in body composition indices as well as maintain the reduced fat mass after training. Thus resistance exercises are recommended as an adjunct for obesity management by reduction in risk factors. Hence, this study is designed to determine the effects of high intensity interval training in combination with resistance exercises verses moderate intensity continuous training on multiple outcome variables including body composition parameters, visceral adiposity, lipid profile and myocardial function in overweight and obese adult population of Pakistan. Afte r obtaining written informed consent from paricipants, they will be screened using 2020 PAR-Q plus and randomly allocated to one of the 2 groups. A self-structured demographic sheet would be employed for recording demographics and required data including the findings of lab investigations. Then participants will be required to undergo all the physical assessment measures such as anthropometric data, 6 minute walk test, lipid profile, body composition analysis and echocardiography. Physical activity levels and QOL would be assessed by filling IPAQ and SF 36 respectively. Exercise training plans would be performed thrice a week on alternate days for a total duration of 10 weeks. All measurements (anthropometric, cardiac, blood and body composition analyses) would be performed at baseline and later after the 10 weeks intervention period. Exercise intensity will be determined by individualized target heart rate zones using Karvonen formula. Strength training intensity will be determined based on 1-RM. Necessary adjustments to speed/grade and resistance will be made over the course of the intervention to ensure that target heart rate zones are achieved at all times. Apart from the exercise programs, a general similar dietary guidance by a nutritionist would also be provided to both of the groups to avoid unhealthy dietary habits.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals categorized as Overweight (BMI 23.0 to 24.9) and Obese-Class I (BMI 25.0 to 29.9).
2. Both males & females willing to participate in the study.
3. Otherwise healthy young adults aged 18-35 and middle-aged adults (36-55 years).
4. No participation in an exercise or PA program during the last 6 months prior to the study.
5. Participants able to complete 6-minute walk test as sub-maximal evaluation test without provoking sign and symptoms.

Exclusion Criteria:

1. Any diagnosed neuromuscular, cardiac, renal, lung, liver disease.
2. Individuals with implantable electrical devices such as pacemakers.
3. Any physical or psychological dysfunction that hinders participation in the study.
4. Individuals already participating in any structured program for weight loss including dietary interventions or usage of nutritional supplements.
5. Individuals unable to complete 6 minute walk test due to any reason (dyspnea, fatigue, chest pain etc).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Body Fat | 10 weeks
  Percentage body fat will be measured using Bioelectrical Impedance Analyzer (Inbody 770) and expressed in forms of percentage (%).
Visceral fat area | 10 weeks
  Visceral fat area will be measured using Bioelectrical Impedance Analyzer (Inbody 770) and expressed in form of centimeter square.

SECONDARY OUTCOMES:
Left Ventricular Mass | 10 weeks
  Left Ventricular Mass depicting myocardial function will be assessed via Echocardiography
Left Ventricular Ejection Fraction | 10 weeks
  Left Ventricular Ejection Fraction depicting myocardial function will be assessed via Echocardiography
Cholesterol/HDL ratio | 10 weeks
  Will be analyzed using Lipid Profile blood testing. A higher score represents poor outcome.
Fat free mass | 10 weeks
  Fat free mass will be measured using Bioelectrical Impedance Analyzer (Inbody 770) and will be expressed in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No